CLINICAL TRIAL: NCT06401733
Title: Metabolic, Inflammatory, Cognitive Risk Stratification, and Intensive Aerobic and Resistance Exercise Intervention for Middle-aged and Older Adults with Type 2 Diabetes Mellitus
Brief Title: Intensive Aerobic and Resistance Exercise Program (IAREP)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Polyclinics, Singapore (Other)
Responsible Party: Principal Investigator, Vivien Xi WU, PhD, Assistant Professor, National University of Singapore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: DSRB-2022/00594
Record Dates: First submitted 2024-04-27; First posted 2024-05-07 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus; Cognitive Impairment; Non-insulin-dependent Diabetes Mellitus; Cognitive Dysfunction
Keywords: T2DM; circuit-based exercise; neurology; dementia; obesity; rehabilitation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction; Dementia; Obesity

STUDY DESIGN:
Intervention Model Description: The study consists of two phases. Phase 1 is a cross-sectional study conducted to gather baseline data and identify eligible participants. Phase 2 involves recruiting participants from the pool established in Phase 1 for an intervention phase. This sequential design allows Phase 1 findings to inform participant selection and eligibility for Phase 2, facilitating a targeted approach to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): 12-week Intensive Aerobic and Resistance Exercise Program (IAREP) intervention group
  Interventions: Other: Intensive Aerobic and Resistance Exercise Program (IAREP)
- Control Group (No Intervention): Subjects that receive their usual care in Jurong polyclinic.

INTERVENTIONS:
Other: Intensive Aerobic and Resistance Exercise Program (IAREP) — IAREP is a combined aerobic exercise and resistance training program that developed by qualified exercise professionals. It encompasses a 12-week exercise intervention, conducted in a blended mode which consists of face-to-face exercise, Zoom exercise, and pre-recorded video exercise.
  Frequency: 3 times exercise per week. Intensity: moderate to vigorous exercise. Time of the exercise: 45-60 mins. Type of exercise: combined aerobic and resistance training.
  Warm-up: aerobic workout with dynamic stretch (for targeted muscles). Aerobic exercise: each session encompasses 5 exercise. Resistance training: each session encompasses 4 exercise, 2 upper body exercise and 2 lower body exercise.
  Cool-down: relax targeted muscles.
  Arms: Intervention Group

SUMMARY:
A 12-weeks Intensive Aerobic and Resistance Exercise Program (IAREP) intervention will be implemented on high-risk and low-risk of cognitive impairment subjects in type 2 Diabetes Mellitus. The study aim to evaluate the effectiveness of IAREP on cognition, metabolic health, physical health, and psychological health in Type 2 Diabetes Mellitus population.

DETAILED DESCRIPTION:
Purpose: A single-site, non-randomized, prospective clinical trial is proposed to determine the significance of an Intensive Aerobic and Resistance Exercise Program on cognitive function, metabolic health, and inflammatory conditions in individuals with Type 2 diabetes mellitus (T2DM) who present with high-risk and low-risk cognitive impairment.

Background and Significance: T2DM is a leading cause of morbidity and mortality among adults worldwide, with approximately 5 million diabetes-related deaths accounting for 12.8% of all-cause mortality in 2015. The prevalence of T2DM in Asia is on the rise, with an anticipated increase from 78 million in 2015 to 140 million by 2040. Asia, therefore, is emerging as the "diabetes epicenter" due to rapid economic development, urbanization, and nutrition transition. T2DM is a complex disease with environmental and genetic contributions that cause many severe complications in middle-aged and older adults, including a higher susceptibility to mild cognitive impairment (MCI) and dementia. The prevalence of cognitive impairment in T2DM ranges from 21.8% to 67.5% worldwide in all adults. Our previous study developed a risk stratification score (RSS) to quickly screen the T2DM population for high-risk or low-risk cognitive impairment. Exercise intervention plays an important role in T2DM management. Aerobic exercise has multiple benefits to metabolic functions, including increasing cardiovascular fitness, improving skeletal muscle capillary density, and reducing body fat. Resistance training is considered a promising intervention for reversing the loss of muscle function and deterioration of muscle structure associated with aging. Intervention strategies, such as the proposed combined aerobic and resistance training program, will provide a guideline to prescribe exercise dosage for individuals with T2DM who are at risk of cognitive impairment.

Methods & Research Plan: The study will recruit 80 subjects, who will be assigned to either the exercise intervention group or the non-exercise control group according to their availability. The intervention group will receive a 12-week Intensive Aerobic and Resistance Exercise Program (IAREP), while the control group will not have IAREP exercise and will continue to receive usual care from Jurong National University Polyclinics. The primary outcomes include cognition, metabolic health, inflammatory conditions, and physical and psychological health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 to 85
* Living in the community
* Diagnosed with type 2 diabetes mellitus (T2DM)
* Literate in English or Mandarin
* Activities of daily living (ADL)-independent
* Obtain at least a score of 5 in short physical performance battery (SPPB) test

Exclusion criteria:

* Severe cognitive (e.g., dementia) or psychiatric disorders (e.g., schizophrenia or severe depression)
* Severe hearing or vision impairments
* Terminally ill medical conditions (e.g., end stage cancer), severe cardiovascular, respiratory (e.g., respiratory failure), or orthopedic conditions (e.g., freeze shoulder)
* Absolute contraindications to aerobic exercise and resistance training programs (e.g., recent myocardial infarction or electrocardiography changes, complete heart block, acute congestive heart failure, unstable angina, uncontrolled hypertension)
* Pregnant or breastfeeding women
* Uncomfortable with video-recording of intervention sessions

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2025-11-04 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function | Baseline and 12 weeks
  Pre- and post-intervention measurements will be conducted. Measure the the change in formal neuropsychological assessment using Vascular Dementia Battery (VDB) for evaluating cognitive function. The neuropsychological assessment covers domains in attention, processing speed, language, visuo-spatial ability, memory and executive function.
Change in metabolic health | Baseline and 12 weeks
  Pre- and post-intervention measurements will be conducted. Measure the change in blood test of HbA1c for metabolic condition.
Change in inflammatory condition | Baseline and 12 weeks
  Pre- and post-intervention measurements will be conducted. Measure the change in blood test of IL6 for inflammatory condition.

SECONDARY OUTCOMES:
Psychological well-beings | 12 weeks
  Post-intervention process evaluation will be conducted from Focus Group Discussion to evaluate the usefulness of the Intensive Aerobic and Resistance Exercise Program (IAREP) intervention.
Change in Short Physical Performance Battery (SPPB) | Baseline and 12 weeks
  Pre- and post-intervention measurements will be conducted. Measure the change in Short Physical Performance Battery (SPPB). The scores range from 0 to 12, higher score means a better outcome.
Change in Body Mass Index (BMI) | Baseline and 12 weeks
  Pre- and post-intervention measurements will be conducted. Measure the change in Body Mass Index (BMI).
Change in sarcopenia condition | Baseline and 12 weeks
  Pre- and post-intervention measurements will be conducted. Measure the change in sarcopenia condition from a rapid sarcopenia screening of Strength, Assistance with walking, Rise from a chair, Climb stairs and Falls (SARC-F). The scores range from 0 to 10, higher score means a worse outcome.
Change in self-care of chronic illness | Baseline and 12 weeks
  Pre- and post-intervention measurements will be conducted. Measure the change in Self-care of Diabetes Inventory. There are 40 items (5 points Likert type) and 4 dimensions: self-care maintenance, self-care monitoring, self-care management and self-care confidence.
Change in health practice behaviour | Baseline and 12 weeks
  Pre- and post-intervention measurements will be conducted. Measure the change in self-perceived ability to implement health-promoting behaviors, which include subscales of Exercise, Nutrition, Responsible Health Practice, and Psychological Well Being. The scores range from 0 to 112, higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Xi Wu, PhD, Principal Investigator — Alice Lee Centre for Nursing Studies, National University of Singapore
Locations (1):
- National University Polyclinic (Jurong Polyclinics), Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No